CLINICAL TRIAL: NCT07291778
Title: The Impact of VeXUS-guided Fluid Management in ICU Populations on Renal Function
Brief Title: VExUS-guided Fluid Management in the ICU
Acronym: VExUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Steven W Fox, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300015346; UAB (Other: UAB)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury; VExUS
Keywords: VExUS; Fluid Management; Acute Kidney Injury; ICU
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain study integrity and minimize bias, multiple layers of blinding will be employed:
  Scanner Blinding: Sonographers performing the VExUS scans are blinded to the patient's randomization status and to all prior scan results. They collect and upload de-identified images labeled only by study ID.
  Interpreter Blinding: The attending physician interpreting the scans (the "overreader") is blinded to randomization status during the image interpretation phase. The overreader reviews both scans for quality and assigns a VExUS score (0-3) before randomization status is revealed.
  Recruiter/Coordinator Role: The research coordinator (unblinded) maintains the randomization list and is responsible for communicating the overread results to the treating team only for patients in the informed arm.
  Primary Team Blinding: For patients in the not-informed arm, the primary clinical team will not receive any VExUS scores or recommendations, and no study-related documentation will be visible in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informed (Experimental): The treating team receives the patient's VExUS results and management recommendations.
  Interventions: Other: Fluid Management
- Non-informed (Placebo Comparator): The treating team remains blinded to all VExUS findings and receives no feedback or recommendations.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Fluid Management — For patients in the informed arm, the overreader will generate standardized recommendations based on the VExUS score:
  VExUS = 0: Recommend a net positive fluid balance.
  VExUS = 1: Recommend a net neutral fluid balance.
  VExUS >= 2: Recommend a net negative fluid balance.
  These recommendations will be communicated to the treating team via a structured process: documentation in the EHR under the POCUS note and verbal handoff to the resident, fellow, and attending on the primary team.
  Arms: Informed
Other: No intervention — Primary team will not be informed about the patient's VExUS score and will not be given recommendations for fluid management
  Arms: Non-informed

SUMMARY:
This study will evaluate the use of the Venous Excess Ultrasound (VExUS) score to guide fluid management in critically ill ICU patients through a prospective, multi-aim design combining observational and randomized components. The study will be conducted in the medical intensive care unit (MICU), multidisciplinary critical care unit (MCCU), and cardiac care unit (CCU) at UAB.

DETAILED DESCRIPTION:
This study will evaluate the use of the Venous Excess Ultrasound (VExUS) score to guide fluid management in critically ill ICU patients through a prospective, multi-aim design combining observational and randomized components. The study will be conducted in the medical intensive care unit (MICU), multidisciplinary critical care unit (MCCU), and cardiac care unit (CCU) at UAB.

Informed Arm: The treating team receives the patient's VExUS results and management recommendations.

Not-Informed Arm: The treating team remains blinded to all VExUS findings and receives no feedback or recommendations.

Each enrolled patient will undergo two VExUS ultrasound assessments:

Timepoint 1 (enrollment): Two scans are performed by separate operators to assess waveform reliability and inter-user reproducibility.

Timepoint 2 (48-72 hours after enrollment): A single scan is performed along with concurrent collection of serum creatinine, intake/output (I&O) balance, and renal replacement therapy (RRT) status.

Each VExUS exam includes Doppler evaluation of the inferior vena cava, hepatic vein, portal vein, renal cortical artery, and renal cortical vein. Scans are saved to secure UAB SharePoint storage labeled with an auto-incrementing study ID.

Blinding Procedures

To maintain study integrity and minimize bias, multiple layers of blinding will be employed:

Scanner Blinding: Sonographers performing the VExUS scans are blinded to the patient's randomization status and to all prior scan results. They collect and upload de-identified images labeled only by study ID.

Interpreter Blinding: The attending physician interpreting the scans (the "overreader") is blinded to randomization status during the image interpretation phase. The overreader reviews both scans for quality and assigns a VExUS score (0-3) before randomization status is revealed.

Recruiter/Coordinator Role: The research coordinator (unblinded) maintains the randomization list and is responsible for communicating the overread results to the treating team only for patients in the informed arm.

Primary Team Blinding: For patients in the not-informed arm, the primary clinical team will not receive any VExUS scores or recommendations, and no study-related documentation will be visible in the electronic health record (EHR).

Statistical Blinding: Data analysts will remain blinded to treatment arm allocation until after all primary outcomes are recorded.

Communication and Clinical Guidance

For patients in the informed arm, the overreader will generate standardized recommendations based on the VExUS score:

VExUS = 0: Recommend a net positive fluid balance.

VExUS = 1: Recommend a net neutral fluid balance.

VExUS >= 2: Recommend a net negative fluid balance.

These recommendations will be communicated to the treating team via a structured process: documentation in the EHR under the POCUS note and verbal handoff to the resident, fellow, and attending on the primary team.

Data Management and Analysis

Two linked data lists will be maintained:

Master List (PHI-protected): Contains patient identifiers and MRNs, stored on a secure UAB server.

Patient Data List (de-identified): Contains study ID, randomization arm, scan quality, interpreter scores, creatinine values, I&O data, RRT status, ICU-free days, hospital-free days, and mortality.

All ultrasound procedures are noninvasive and adhere to ACEP emergency ultrasound standards. Protected health information will remain secured on institutional servers, and only de-identified data will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Admitted to the MICU, MCCU, or CCU within 24 hours of admission
* Acute kidney injury (AKI) (based on Kidney Disease: Improving Global Outcomes (KDIGO) criteria)
* Adequate acoustic windows for a complete VExUS scan

Exclusion Criteria:

* < 18 years old
* pregnant women
* End-stage renal disease (ESRD) or prior renal transplant
* Acute tubular necrosis (ATN) defined by urinalysis (≥2+ protein, ≥2+ blood, ≥1 muddy brown cast, ≥1 RBC cast, or ≥1 dysmorphic RBC)'
* Prior Whipple procedures
* currently incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital Mortality | up to 30 days
  In-hospital mortality: Death from any cause before hospital discharge, within the 30-day window.
Renal Replacement Therapy | up to 30 days
  New receipt of Renal Replacement Therapy (RRT): Receiving dialysis or another form of RRT for the first time.
Persistent Renal Dysfunction | up to 30 days
  Persistent renal dysfunction: The final serum creatinine value before hospital discharge (within 30 days) is 200% (twice) or more of the patient's baseline creatinine value.
Creatinine Change | 48 - 72 hrs
  A patient's change in creatinine from enrollment at the 48 - 72 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham Medical Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided